CLINICAL TRIAL: NCT05640297
Title: "Impact of Kangaroo Mother Care Plus Massage Therapy on Growth of Preterm Low Birth Weight Infants at Discharge"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Collaborators: Bangladesh College Of Physicians And Surgeons (BCPS) (Other)
Responsible Party: Principal Investigator, Dr. Sonia Aktar, Doctor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3838
Record Dates: First submitted 2022-11-15; First posted 2022-12-07 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Weight Gain
MeSH Terms: conditions — Weight Gain | interventions — Massage

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KMC with Massage therapy (Experimental): Preterm low birth weight babies who will get KMC will also receive massage therapy
  Interventions: Behavioral: KMC with Massage therapy
- KMC only (No Intervention): Preterm low birth weight babies who will get KMC only

INTERVENTIONS:
Behavioral: KMC with Massage therapy — investigator will provide tactile and kinesthetic massage
  Arms: KMC with Massage therapy

SUMMARY:
Kangaroo mother care plus massage therapy will lead to improved growth of preterm low birth weight infants at discharge.

DETAILED DESCRIPTION:
Primary phase of the transition from the fetal to post-natal period is the most important, vulnerable and stressful phase in human life. Hence, care methods that facilitate better adaptation of neonates with early post¬natal environment have an important role in growth of newborns. Attachment is a unique relationship between the parents and their infants that begins during pregnancy when fetus grows in uterus and continues to the postnatal period with the relationship of mother and baby. This reciprocal parent-infant relationship is an essential element of the attachment process that helps relaxation of both mother and the infant. Kangaroo mother care has facilitated infant growth and decreased morbidities and hospital stay. Adding massage therapy may potentiate the kangaroo mother care benefits and better growth in preterm low birth weight infants admitted in neonatal intensive care unit. However, there is a very few published studies from Bangladesh regarding this. The objective of this study is to evaluate whether kangaroo mother care plus massage therapy is associated with better growth of preterm low birth weight infants.

This study will be conducted in the department of Neonatology in Bangabandhu Sheikh Mujib Medical University over a period of eighteen months. After detailed history taking and thorough general and systemic examination the newborn will enter in to intervention or control group after taking informed written consent. Randomization will be done by random allocation software (version 2.0 developed by Mahmood Saghaei, Iran). Patient will be enrolled according to the inclusion and exclusion criteria. Thereafter control group will receive standard kangaroo mother care and intervention group will get massage therapy along with kangaroo mother care, up to discharge both group will be meticulously monitored by the investigator. Data will be collected by structured questionnaire and analysis will be done by The Statistical Package for Social Sciences (SPSS), version 25.

ELIGIBILITY:
Inclusion Criteria:

* 1. Gestational age <34 weeks. or 2. Neonates weighing less than 2000 gm. With any one of the following

  1. Hemodynamically stable.
  2. Preterm neonate with up to 2 L/min O2 support by nasal canula or prong.

Exclusion Criteria:

* Inclusion Criteria:

  1. Gestational age <34 weeks. or
  2. Neonates weighing less than 2000 gm. With any one of the following

     1. Hemodynamically stable.
     2. Preterm neonate with up to 2 L/min O2 support by nasal canula or prong.

Exclusion Criteria:

1. Hemodynamically unstable critically ill neonates.
2. Newborn with severe perinatal asphyxia and seizure
3. Newborn requiring exchange transfusion.
4. Newborn with major congenital and chromosomal abnormalities.
5. Newborn with sepsis, IVH, shock, necrotizing enterocolitis.
6. Newborn with major surgical illness.

Ages: 1 Hour to 28 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Weight in grams | 18 months
  Pattern of weight gain in grams using KINLEE EBST-20 weighing scale.

SECONDARY OUTCOMES:
OFC in centimeter | 18 months
  pattern of head growth using measuring tape

OTHER OUTCOMES:
length of hospital stay in days | 18 months
  to see how many days the baby needs hospital care

CONTACTS AND LOCATIONS:
Overall Officials: sonia aktar, MBBS,DCH, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- BSMMU, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
After completion principle investigator will share
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: december,2022